CLINICAL TRIAL: NCT04898075
Title: Quit Nicotine: E-Cig Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000028718; 20YVNR35460041 (Other: American Heart Association)
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: E-Cig Use
Keywords: Contingency management
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Contingency Management (CM) for nicotine abstinence (Experimental): Participants will be paid increasing amounts of payment for each negative saliva cotinine test.
  Interventions: Behavioral: Remote Contingency Management (CM) for nicotine abstinence
- Control (Placebo Comparator): Participants will be paid for providing saliva nicotine test, regardless of whether the test is positive or negative.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Remote Contingency Management (CM) for nicotine abstinence — Participants will be paid increasing amounts of payment for each negative saliva cotinine test.
  Arms: Remote Contingency Management (CM) for nicotine abstinence
Other: Control — Participants will be paid for providing saliva nicotine test, regardless of whether the test is positive or negative.
  Arms: Control

SUMMARY:
The purpose of this study is to find out if a new intervention helps teenagers who vape nicotine quit vaping. The program involves two parts: giving rewards (also called contingency management [CM]) and online video counseling (also called cognitive behavioral therapy [CBT]).

DETAILED DESCRIPTION:
Eligible participants will participate in a 4-week long Remote Contingency Management (Remote CM) intervention that involves the delivery of CM procedures using tablets, weekly vaping cessation CBT sessions, and follow-up appointments at 1, 3, 6, and 12 months.

Aim 1. To examine the feasibility, acceptability, and efficacy of web-based, remote Contingency Management (CM) for nicotine abstinence plus individualized Cognitive Behavioral Therapy (CBT) among youth e-cigarette (e-cig) users. High school students 13-19 years old who are regular e-cig users who want to quit (N=100) will be randomized to the Active group (CM for nicotine abstinence; reinforcement for negative saliva nicotine/cotinine; n=50) or Control group (reinforcement for providing saliva nicotine; n=50) for 4 weeks. Both groups will receive weekly CBT during this time (2 sessions prior to quitting, 4 weekly sessions after quitting). The investigators expect the Active group to have better treatment outcomes (7-day point prevalence abstinence at end-of-treatment [EOT] and follow ups [1, 3, 6, and 12- months]) than the Control group.

Aim 2. To examine the relationship between e-cig use characteristics, dependence, e-cig withdrawal, and treatment outcome/abstinence. It is anticipated that using higher nicotine concentrations; using a greater total number of flavors; vaping frequently or endorsing habitual use; and reporting fewer prior quit attempts will be associated with experiencing more severe dependence and e-cig withdrawal. In turn, researchers expect that experiencing more severe e-cig dependence before quitting and/or more severe withdrawal following the quit date will predict treatment failure (e.g., failure to achieve abstinence, a longer duration until abstinence is achieved, higher cotinine levels)

Aim 3. To test for changes in neurocognitive functioning in adolescent e-cig users across treatment for e- cig cessation. In this study, the Adolescent Brain and Cognitive Development study neurocognitive battery will be utilized. This will be administered at baseline and end of treatment to all participants (N=100). It is anticipated that youth e-cig users will show improvements in neurocognitive task performance (e.g., working memory, attention) from baseline to end of treatment. It is also predicted that improvements in neurocognitive task performance will be related to abstinence from e-cigs during treatment

ELIGIBILITY:
Inclusion Criteria:

* High school students between ages 13-20 years (plus 5 high school aged pilot participants)
* Able to read and write
* Regular e-cig users using nicotine (primary e-cig users with or without other tobacco use who report using e-cigs at least 4 days/week and have urine cotinine levels ≥200 ng/ml as determined by 1 Panel Quickscreen Cotinine/Nicotine Test Dipcard, COT200; Countrywide Testing) who want to quit. A repeat urine may be tested with the 200ng/ml dip test if subject reports levels of vaping that may be consistent with higher levels of cotinine.
* Does not meeting criteria for dependence on other psychoactive substances, psychosis, major depression or panic disorder based on psychological evaluation.

Exclusion Criteria:

* Currently enrolled in, or planning to enroll in any other behavioral or pharmacological treatments for cessation of nicotine or vaping.
* Current criteria for Substance Use Dependence (SUD) on other psychoactive substances. Endorsement of mild Cannabis Use Disorder will be allowed, due to the fact than many nicotine users may also be vaping cannabis
* Current diagnosis of psychosis or evidence of significant homicidal/suicidal risk.
* Current diagnosis of a significant mental health disorder that is not being treated by a mental health practitioner with either behavioral and/or pharmacological interventions.
* Regular use of any psychoactive drugs including anxiolytics and antidepressants unless the adolescent has been taking the medication consistently for 2 months, the medication is currently being monitored by a physician, and the condition for which the medication is taken is considered to be stable.
* Females who report being pregnant or lactating

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Change in 7-day point prevalence abstinence | End of treatment at week 4, 1, 3, 6, and 12 month
  Self reported of no e-cig usage during the 7 days prior and confirmed negativity with cotinine levels of 30ng/mL (Alere iScreen OFD Cotinine Saliva Test; Countrywide Testing).

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No